CLINICAL TRIAL: NCT04478760
Title: Reference Intervals for 27 Routine Chemistry and Immunoassay Tests in Transgender Adults on Stable Hormone Therapy
Brief Title: Trans & Non-binary Reference Intervals While on Hormone Therapy Study
Acronym: TransRIHTS
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TransRIHTS Protocol
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Transgender Persons; Hormone Replacement Therapy; Reference Values

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Masculinising therapy: Healthy transgender (including non-binary) adults who are on testosterone-containing hormone therapies.
- Feminising therapy: Healthy transgender (including non-binary) adults who are on oestrogen-containing hormone therapies.

SUMMARY:
This study will find out what the reference intervals are for common blood tests in transgender people taking hormone therapy.

Reference intervals help doctors interpret blood test results. They are expressed as two numbers, and most normal results fall between them. If a results fall outside of them, it may be because of a disease. Some blood tests are also affected by normal difference between people, such as age, sex or ethnicity. For these tests, different reference intervals are given for each group of people. Having accurate reference intervals benefits patients because it allows doctors to identify disease faster.

Transgender people have a gender identity which does not match their sex characteristics at birth. Gender identity is the feeling of being a gender, and sex is the biological aspects of growing up male or female. Transgender people may use hormone therapy to help change their appearance to fit their gender identity. This involves taking either oestrogen or testosterone.

For blood tests which are affected by sex, it is not clear what reference intervals should be used for transgender people who are on hormone therapy. This is because they have a mixture of male and female sex characteristics. Answering this question will allow doctors to identify disease in them faster.

The study will take place at cliniQ, at King's College Hospital, which provides health services to transgender people. It will recruit healthy transgender people who attend the clinic for blood tests to monitor their hormone therapy. Participants will fill out a questionnaire, give a urine sample, then have their appointment as normal. Extra tests will also be performed on their blood sample. The aim is to recruit 240 participants. Participant's tests results will then be used to calculate reference intervals.

The study is funded by Viapath Group LLP.

ELIGIBILITY:
Inclusion Criteria:

* Transgender or nonbinary people.
* Aged 18 or older.
* Taking testosterone or oestrogen therapy.
* For 12 months or more.
* Having routine hormone therapy monitoring at the clinic.

Exclusion Criteria:

* Unable to give informed consent (including participants who cannot communicate in English).
* History of chronic liver disease, chronic kidney disease, diabetes, or severe cardiovascular disease (including myocardial infection, deep vein thrombosis, stroke and pulmonary embolism).
* Blood test results that indicate severe disease.
* Pregnant or within one year after childbirth.
* Other conditions which could put participants at risk by participating, or which could influence the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are eligible if they are transgender, that is, their gender is different from their sex assigned at birth.
Study Population: Healthy transgender adults who have been taking masculinising for feminising hormone therapy for at least 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Reference interval for transgender patients on hormone therapy | 1 day
  Establish reference intervals for routine chemistry and immunoassay test for transgender people on hormone therapy. Establish separate reference intervals for people on masculinising and feminising therapy if they differ substantially.

SECONDARY OUTCOMES:
Compare the reference intervals in patients taking different hormone therapy formulations. | 1 day
  Compare different hormone therapy formulations to establish whether there are clinically significant difference in their effects on reference intervals.
Compare transgender reference intervals to the existing ones | 1 day
  Compare the reference values for transgender people on hormone therapy with the existing cisgender reference intervals to establish whether they are similar enough for the cisgender reference intervals to be used instead.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brady, FRCP, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- Caldecot Centre, King's College Hospital, 15-22 Caldecot Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, deidentified participant-level data and the analysis files will be uploaded to an open access repository within 6 months of the publication of the findings.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within 6 months of the publication of the results of the research.
Access Criteria: Public access to deidentified data.